CLINICAL TRIAL: NCT00945568
Title: Preoperative Oral Supplementation With Carbohydrate and Branched-chain Amino Acid-enriched Nutrient Improves Postoperative Quality of Life in Patients Undergoing a Hepatectomy
Brief Title: Preoperative Oral Supplementation With Branched-Chain Amino Acids (BCAA) Improves Postoperative Quality of Life
Acronym: KMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kochi University (Other)
Responsible Party: Kochi Medical School, Kochi University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AEN-0901; KMS
Record Dates: First submitted 2009-07-14; First posted 2009-07-24 (Estimated); Last update posted 2009-07-24 (Estimated); Status verified 2009-07

CONDITIONS: Hepatocellular Carcinoma; Chronic Liver Disease
Keywords: QOL; liver
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aminolaban EN (Experimental): Aminoleban EN™ was administered at a dose of 100 g per day commencing two weeks prior to surgery. A 100 g dose of Aminoleban EN™ contains 13.0 g of free amino acids, 13.0 g of gelatin hydrolysate, 1.0 g of casein, 62.1 g of carbohydrate, 7.0 g of lipid, glycyrrhizin, and other components, producing 420 kcal. The AEN group included 40 patients who were administered 100 g of Aminoleban EN™ as 50 g during the day and 50 g as a late evening snack.
  Interventions: Drug: Aminoleban EN
- Control (No Intervention): The patients were divided into two groups including one group administered Aminoleban (the AEN group) and a control group given no additional dietary supplementation. The total caloric energy intake per day during the study period was assumed to be equal to Aminolaban EN group.
  Interventions: Drug: Aminoleban EN

INTERVENTIONS:
Drug: Aminoleban EN — benefits of this drug for patients who undergoing liver resection for HCC
  Other Names: AEN

SUMMARY:
The aims of this study are (1) to study the benefit of branched-chain amino acids enriched nutrient-mixture by analyzing a variety of clinical parameter, including laboratory data, the duration of hospitalization after the surgery, and (2) To investigate the postoperative quality of life (QOL) in receiving peri-operatively branched-chain amino acids enriched nutrient-mixture in patients who undergone the hepatic management for hepatocellular carcinoma (HCC) with chronic liver disease.

DETAILED DESCRIPTION:
Patients with cirrhosis of the liver complicated with HCC are often in a state of protein energy malnutrition. A limited number of studies have indicated an important role for nutritional support in the surgical management of patients who have undergone hepatic resection for HCC. In a preliminary study, we reported the clinical efficacy of supplementation with branched-chain amino acids in a small number of patients with liver cirrhosis who underwent hepatic surgery for HCC. The aims of this study are (1) to study the benefit of branched-chain amino acids enriched nutrient-mixture by analyzing a variety of clinical parameter, including laboratory data, the duration of hospitalization after the surgery, and (2) To investigate the postoperative QOL in receiving peri-operatively branched-chain amino acids enriched nutrient-mixture in patients who undergone the hepatic management for HCC with chronic liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent elective liver resection for the treatment of hepatocellular carcinoma or adenocarcinoma with chronic liver diseases.

Exclusion Criteria:

* Body weight loss greater than 10 per cent during the 6 months prior to surgery,
* The presence of distant metastases, or seriously impaired function of vital organs due to respiratory, renal or heart disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To study the benefit of branched-chain amino acids enriched nutrient-mixture by analyzing a variety of clinical parameter, including laboratory data, the duration of hospitalization after the surgery. | 3-6 months

SECONDARY OUTCOMES:
To investigate the safety, rationality and postoperative QOL in receiving peri-operatively branched-chain amino acids enriched nutrient-mixture in patients who undergone the hepatic management for HCC with chronic liver disease. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kazuhiro Hanazaki, Prof, Study Director — Kochi University
Locations (2):
- Japan (2):
  - Kochi Medical School, Nankoku, Kochi
  - Kochi Medical School, Kochi University, Nankoku, Kohasu-Okocho

REFERENCES:
- [Derived] Okabayashi T, Iyoki M, Sugimoto T, Kobayashi M, Hanazaki K. Oral supplementation with carbohydrate- and branched-chain amino acid-enriched nutrients improves postoperative quality of life in patients undergoing hepatic resection. Amino Acids. 2011 Apr;40(4):1213-20. doi: 10.1007/s00726-010-0748-3. Epub 2010 Sep 18. PMID 20852905